CLINICAL TRIAL: NCT00734292
Title: A Randomized, Placebo-controlled, Double-blind, Crossover, Single-dose Exposure Study to Evaluate the Early Bronchodilating Effect of FlutiForm 100/10 µg HFA pMDI and FlutiForm 250/10 µg HFA pMDI, Compared to Placebo in Adult Subjects With Mild to Moderate Asthma
Brief Title: Single-dose Crossover Study to Evaluate the Early Bronchodilating Effect of FlutiForm HFA pMDI in Adult Subjects With Mild to Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SkyePharma AG (Industry)
Collaborators: Abbott (Industry)
Responsible Party: SkyePharma AG, SkyePharma AG
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SKY2028-2-002
Record Dates: First submitted 2008-08-04; First posted 2008-08-14 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Mild to Moderate Asthma
Keywords: Asthma; Asthma Mild to Moderate
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Formoterol Fumarate; fluticasone-formoterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- I (Placebo Comparator): * Period 1 Treatment Regimen A: FlutiForm 250/10 ug
  * Period 2 Treatment Regimen B: FlutiForm 100/10 ug
  * Period 3 Treatment Regimen C: placebo
  Interventions: Drug: fluticasone propionate, formoterol fumarate
- II (Placebo Comparator): * Period 1 Treatment Regimen B: FlutiForm 100/10 ug
  * Period 2 Treatment Regimen C: placebo
  * Period 3 Treatment Regimen A: FlutiForm 250/10 ug
  Interventions: Other: fluticasone propionate, formoterol fumarate
- III (Placebo Comparator): * Period 1 Treatment Regimen C: placebo
  * Period 2 Treatment Regimen A: FlutiForm 250/10 ug
  * Period 3 Treatment Regimen B: FlutiForm 100/10 ug
  Interventions: Other: fluticasone propionate, formoterol fumarate

INTERVENTIONS:
Drug: fluticasone propionate, formoterol fumarate — ● Period 1 Treatment Regimen A: FlutiForm 250/10 ug
  FlutiForm HFA pMDI (250/10 ug); (two actuations of FlutiForm HFA pMDI 125/5 ug/actuation)
  ● Period 2 Treatment Regimen B: FlutiForm 100/10 ug
  FlutiForm HFA pMDI (100/10 ug); (two actuations of FlutiForm HFA pMDI 50/5 ug/actuation)
  ● Period 3 Treatment Regimen C: placebo
  SKP placebo; (two actuations)
  Other Names: FlutiForm
  Arms: I
Other: fluticasone propionate, formoterol fumarate — ● Period 1 Treatment Regimen B: FlutiForm 100/10 ug
  FlutiForm HFA pMDI (100/10 ug); (two actuations of FlutiForm HFA pMDI 50/5 ug/actuation)
  ● Period 2 Treatment Regimen C: placebo
  SKP placebo; (two actuations)
  ● Period 3 Treatment Regimen A: FlutiForm 250/10 ug
  FlutiForm HFA pMDI (250/10 ug); (two actuations of FlutiForm HFA pMDI 125/5 ug/actuation)
  Other Names: FlutiForm
  Arms: II
Other: fluticasone propionate, formoterol fumarate — ● Period 1 Treatment Regimen C: placebo
  SKP placebo; (two actuations)
  ● Period 2 Treatment Regimen A: FlutiForm 250/10 ug
  FlutiForm HFA pMDI (250/10 ug); (two actuations of FlutiForm HFA pMDI 125/5 ug/actuation)
  ● Period 3 Treatment Regimen B: FlutiForm 100/10 ug
  FlutiForm HFA pMDI (100/10 ug); (two actuations of FlutiForm HFA pMDI 50/5 ug/actuation)
  Other Names: FlutiForm
  Arms: III

SUMMARY:
The primary purpose of this study is to evaluate the early bronchodilating effect of SKP FlutiForm HFA pMDI compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented history of mild to moderate asthma currently taking a stable dose of inhaled corticosteroid

Exclusion Criteria:

* Participation in a prior FlutiForm study
* Smoking history within the last 12 months,
* Significant, non-reversible, pulmonary disease
* Life-threatening asthma within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline FEV1 to post study drug dosing FEV1 | 3 minutes

SECONDARY OUTCOMES:
Change from baseline FEV1 to post study drug dosing FEV1 | 8, 15, 30, and 60 minutes

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Investigational Site, Anaheim, California
  - Investigational Site, Mission Viejo, California
  - Investigational Site, Denver, Colorado
  - Investigational Site, Valrico, Florida
  - Investigational Site, Medford, Oregon
  - Investigational Site, Portland, Oregon
  - Investigational Site, Richmond, Virginia
  - Investigational Site, West Allis, Wisconsin